CLINICAL TRIAL: NCT03230565
Title: A Prospective Comparison of Pain and Analgesia in Patients With Continuous Peripheral Nerve Block Catheters Using Continuous Infusion or Scheduled Bolus Infusion
Brief Title: Continuous Infusions vs Scheduled Bolus Infusions
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jean-Louis Horn, Professor of Anesthesiology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 41434
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Surgical Procedure, Unspecified; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Comparison of two groups: 1) Continuous infusion group 2) Bolus infusion group
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Investigators and participants will be masked to treatment group. Care providers will be necessarily unmasked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Continuous Infusion (Active Comparator): Local anesthetic medication (Ropivacaine 0.2%) is provided at a continuous basal rate.
  Interventions: Drug: Ropivacaine
- Intermittent Bolus Infusion (Active Comparator): Local anesthetic medication (Ropivacaine 0.2%) is provided in scheduled, intermittent boluses.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Patient will be given a continuous infusion of local anesthetic.
  Other Names: Continuous infusion
  Arms: Continuous Infusion
Drug: Ropivacaine — Patient will be given a scheduled intermittent bolus of local anesthetic.
  Other Names: Bolus Infusion
  Arms: Intermittent Bolus Infusion

SUMMARY:
The goal of the study is to compare continuous infusions and scheduled bolus infusions for peripheral nerve blocks and their effect on post-surgical pain.

DETAILED DESCRIPTION:
Regional anesthetic techniques are an integral part to many anesthetic approaches, providing both intraoperative and postoperative anesthesia and analgesia. Regional anesthesia peripheral nerve blocks have been shown to reduce postoperative pain and improve measures such as opioid requirements and readiness for discharge. By using a catheter technique for continuous peripheral nerve blocks, analgesia can be extended well into post-operative days 2 and 3, further extending these benefits. Historically these catheters have implemented a continuous dosing regimen of local anesthetic, but increasingly there is evidence of improved analgesic outcomes without adverse effects by using a scheduled bolus dosing regimen. Many institutions have implemented this new protocol for catheter dosing. The beneficial effect of scheduled bolus dosing has not been studied in all blocks and all surgical procedures.

The study will consist of three independent arms, each designed to evaluate a different nerve block site: interscalene, adductor canal, and infraclavicular. A total of 60 patients will be enrolled in each arm.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients presenting for nerve block catheters for post-operative analgesia
* ASA physical status I, II, or III.

Exclusion Criteria:

* Pregnancy
* Incarceration
* Age <18
* BMI >35
* Pre-operative opioid use >30 mg morphine equivalents per day
* Inability to communicate with investigators by telephone
* Pre-existing neuropathy of the operative extremity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Post-surgical pain | Post-operative day 0, 1, and 2
  Pain scores will be collected using a Numeric Rating Scale (NRS) from 0-10, where 0 is the lowest and 10 is the highest pain level.

SECONDARY OUTCOMES:
Opioid consumption | Post-operative day 0, 1, and 2
  The amount of opioid analgesics (converted to total morphine milligram equivalents) taken by patients will be recorded.
Local anesthetic use | Post-operative day 1 and 2
  The amount of supplemental local anesthetic boluses self-administered by patients will be recorded (in mL).
Quality of recovery | Post-operative day 1 and 2
  Quality of recovery will be assessed using a Quality of Recovery (QoR-15) questionnaire. The QoR15 scores range from 0 to 150, where 0 is poor recovery and 150 is excellent recovery.
Evidence of diaphragmatic paralysis | Post-operative day 1 and 2
  Ability to breathe will be assessed as a part of QoR-15 questionnaire on 11-point scale, where 0 is never being able to breathe easily and 10 is always being able to breathe easily.
Patient satisfaction | Post-operative day 1 and 2
  Patients will be asked to assess their satisfaction with pain management (Yes/No).

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis-Horn, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No